CLINICAL TRIAL: NCT00217464
Title: Multicenter Study of Fulvestrant (Faslodex®) in Early, Recurrent Prostate Cancer Following Local Therapy: A Phase II Trial
Brief Title: Fulvestrant in Treating Patients With Recurrent Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed for futility
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441210; RPCI-I-17203; ZENECA-IRUSFULV0026
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fulvestrant (Experimental): Fulvestrant will be provided as 250 mg in 5 mL as a pre-tilled syringe. Fulvestrant will be administered as 500 mg, that is, 2 injections of 5 mL, one into each buttock im on day 0. A single 250 mg in 5 mL injection will be administered on day 14 followed by a single 250 mg in 5 mL dose on day 28 and monthly thereafter.
  Interventions: Drug: fulvestrant

INTERVENTIONS:
Drug: fulvestrant — intramuscularly

SUMMARY:
RATIONALE: Estrogen may cause the growth of prostate cancer cells. Hormone therapy using fulvestrant may fight prostate cancer by blocking the use of estrogen by the tumor cells.

PURPOSE: This phase II trial is studying how well fulvestrant works in treating patients with recurrent prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether fulvestrant can slow the rise of prostrate-specific antigen (PSA) level in patients with early recurrent adenocarcinoma of the prostate after radical prostatectomy or irradiation.

Secondary

* Determine the utility of monitoring serum PSA in patients treated with this drug.
* Determine the safety of this drug in these patients.
* Determine changes in bone mineral density and markers of bone resorption in patients with PSA-only failure treated with this drug.

OUTLINE: This is an open-label, single group assignment study.

Patients receive fulvestrant intramuscularly on days 0, 14, and 28. Treatment repeats once a month in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 32 patients will be accrued for this study for 84 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Early recurrent disease, defined by 1 of the following criteria:

    * Prostate-specific antigen (PSA) ≥ 2.0 ng/mL AND clearly rising within the past 3 months for patients who underwent prior prostatectomy with or without radiotherapy
    * PSA ≥ 4.0 ng/mL AND clearly rising from the lowest value obtained within the past 6 months for patients who underwent prior definitive radiotherapy only
* No evidence of clinical recurrence,* as defined by the following criteria:

  * Digital rectal exam negative
  * No local recurrence by CT scan or MRI of the pelvis
  * No evidence of bone metastasis by bone scan NOTE: *Prostascint scan results are not considered evidence of recurrence
* Underwent prior curative treatment comprising radical prostatectomy with or without adjuvant radiotherapy OR definitive radiotherapy alone
* Testosterone (total or free) > than lower limit of normal

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC > 3,500/mm^3
* Platelet count > 100,000/mm^3
* No history of bleeding diathesis

Hepatic

* INR < 1.6
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT or AST ≤ 2.5 times ULN
* No severe hepatic impairment that would preclude study participation or compliance

Renal

* Creatinine ≤ 2.0 mg/dL
* No severe renal impairment that would preclude study participation or compliance

Cardiovascular

* No unstable or uncompensated cardiac condition that would preclude study participation or compliance

Pulmonary

* No unstable or uncompensated respiratory condition that would preclude study participation or compliance

Other

* No history of hypersensitivity to active or inactive excipients of fulvestrant (e.g., castor oil)
* No other severe condition that would preclude study compliance (e.g., abuse of alcohol or drugs or psychotic states) or participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* More than 6 months since prior neoadjuvant or adjuvant androgen deprivation therapy or luteinizing hormone-releasing hormone antagonist therapy
* No other prior or concurrent hormonal therapy

Radiotherapy

* See Disease Characteristics
* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* More than 4 weeks since prior experimental drug treatment
* No concurrent anticoagulant therapy except antiplatelet therapy
* No other concurrent therapy for prostate cancer
* No other concurrent therapy known or suspected of altering androgen metabolism or androgen levels

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-06; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald L. Trump, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fulvestrant: Patients receive fulvestrant intramuscularly on days 0, 14, and 28. Treatment repeats once a month in the absence of disease progression or unacceptable toxicity.
  fulvestrant: intramuscularly
Period: Overall Study
Arm/Group | Fulvestrant
Started | 17
Completed | 0
Not Completed | 17
Not completed — Progression | 15
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Fulvestrant
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.01 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Respond to Treatment.
Description: Response is defined to be the clear slowing of the rate of increase of PSA levels with time
Time Frame: 90, 60, and 30 days pre-treatment, the day of start therapy (day 0) and 30, 60 and 90 days post-treatment
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fulvestrant
Number analyzed (Participants) | 17
percentage of participants | 0 [0 to 18.4]

2. Secondary Outcome: Number of Participants With Progressive Disease at Day +90
Description: Progressive Disease is defined as failure to achieve a statistically significant decrease in PSA rise after the day +90 PSA value
Time Frame: 90, 60, and 30 days pre-treatment, the day of start therapy (day 0) and 30, 60 and 90 days post-treatment
Population: All treated and eligible patients
Measure: Number; unit: participants
Arm/Group | Fulvestrant
Number analyzed (Participants) | 17
participants | 15

ADVERSE EVENTS:
Arm/Group | Fulvestrant
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant (N=17)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Injection site inflammation (General disorders) | 1 (1)
Injection site pain (General disorders) | 9 (9)
Injection site reaction (General disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (6)
Hypernatraemia (Metabolism and nutrition disorders) | 4 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hot flush (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes